CLINICAL TRIAL: NCT04182477
Title: The Impact of Age and Number of Previous Anesthesia on the Development of Mild Cognitive Decline (MCI) in Patients Enrolled for Cardiac Surgery
Brief Title: Age and Number of Previous Anesthesia on the Development of Mild Cognitive Decline (MCI)
Acronym: MCI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: Eleonora Maran (Unknown); Alessandro de Laurenzis (Unknown)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal investigator, University of Padova
Other Study IDs: ZivagoMCI
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with at least one general anesthesia in anamnesis: Patients who underwent during their life at least one anesthesia in anamnesis
  Interventions: Diagnostic Test: Montreal Cognitive Assessment
- Patient without general anesthesia in anamnesis: Patients who never underwent general anesthesia during their life
  Interventions: Diagnostic Test: Montreal Cognitive Assessment

INTERVENTIONS:
Diagnostic Test: Montreal Cognitive Assessment — Neuro-cognitive test evaluating general mental status and performance
  Other Names: MoCA

SUMMARY:
Mild Cognitive Impairment (MCI), diagnosed with Montreal Cognitive assessment test (MoCA) define a condition that is insufficient to meet the threshold for a diagnosis of dementia, and it is an increasing health problem.

It has been related to age and comorbilities, but the linkage between MCI and number of previous anesthesia is still unclear.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is a common neuropsychiatric term encompassing a greater-than-expected cognitive decline for patient's age and schooling and no more than mild functional impairment that is insufficient to meet the threshold for a diagnosis of dementia (DSM-V: "mild neurocognitive disorder") thus forming part of a declining cognitive trajectory.

For the diagnosis of MCI, the core clinical criteria are: concern about a change in cognition, impairment in one or more cognitive domains, preservation of independence in functional abilities and no presence of dementia.

The Montreal Cognitive Assessment (MoCA), a test that was developed specifically for detection of MCI, has a sensitivity of 80 to 100% and specificity of 50 to 76% using a cut-off point of 25 to make diagnosis, and it has been suggested that it is better than Mini Mental Status Evaluation (MMSE) in accurately differentiating individuals with MCI from those with normal cognition.

Various risk factors have been proposed for MCI, in particular the role of multiple biological, behavioural, social and environmental factors have been investigated.

Of them, increasing in age, lower educational level, sleep-disordered breathing and vascular risk factors (e.g. diabetes and hypertension) seem to be the most important.

It has been estimated that MCI is itself a risk factor both for dementia (it converts to dementia at a rate of 10% per year, for delirium and Post-Operative Cognitive Decline (POCD).

Hence, this study aims to investigate the incidence of MCI in cardiac-surgery adult patients, enlisted for Coronary Artery By-Pass Grafting (CABG) or Valve Surgery, and to investigate the role of previous general anaesthesia in anamnesis as a risk factor for MCI evenience.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing Cardiac - Surgery intervention with extracorporeal circulation

Exclusion Criteria:

* Neurological disease before surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective Observational Case-Control
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Mild cognitive impairment (MCI)in patients enrolled for Cardiac Surgery | Patients will be subjected to Montreal Cognitive Assessment (MOCA) test one day before surgery. T
  Patients will be interviewed by a psychologist assessing diagnosis of MCI with Montreal Cognitive Test (Better performance with higher scores)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Italy